CLINICAL TRIAL: NCT00222170
Title: Esophagoprotection by Rabeprazole Mediated by Restoration of an Impairment in Esophageal Mucin Production: Its Potential Therapeutic Benefit in Patients With Gastroesophageal Reflux Disease (GERD)
Brief Title: Rabeprazole in Subjects With Gastroesophageal Reflux Disease (GERD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kansas (Other)
Collaborators: PriCara, Unit of Ortho-McNeil, Inc. (Industry); Eisai Inc. (Industry)
Organization: University of Kansas Medical Center (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RE Study
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2009-05-08 (Estimated); Status verified 2007-08

CONDITIONS: Esophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Rabeprazole

SUMMARY:
The purpose of this study is to determine the production of mucin in GERD/RE subjects before and after 8 weeks of treatment with rabeprazole.

DETAILED DESCRIPTION:
Enrolled patients will undergo collection of salivary and esophageal secretions. Subsequently, all patients will receive rabeprazole (20mg QD) for 8 weeks and will be re-endoscoped to confirm complete healing of reflux esophagitis. In patients with completely healed reflux esophagitis the second collection of salivary and esophageal secretion will be implemented. In both secretions, adequately coded for the laboratory Research Fellow (blinded in terms of which sample is collected before and which after treatment with rabeprazole) the content of mucin will be measured using commercially available assay and its secretion expressed in units per minute of collection time.

ELIGIBILITY:
Inclusion criteria: 24 patients with endoscopically confirmed reflux esophagitis (Grades A-D according to LA classification) in patients with chronic symptoms of GERD (heartburn with or without regurgitation) between the age of 19 and 79, 12M & 12F, will be included.

Exclusion criteria: History of GI surgery, primary esophageal motor disorders, any systemic disease, history of drug or alcohol abuse, pregnancy or nursing, allergy to the same drug class as rabeprazole, the need for any concurrent therapy that affects salivary secretion (causing so-called "dry mouth syndrome").

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-05; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Measure of concentration and output of esophageal mucus in esophageal secretion before and after 8 weeks of therapy with rabeprazole

SECONDARY OUTCOMES:
Esophageal mucin measurement comparisons on samples collected before and after rabeprazole therapy

CONTACTS AND LOCATIONS:
Overall Officials: Jerzy Sarosiek, PhD, Principal Investigator — University of Kansas Medical Center; Mojtaba S. Olyaee, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States